CLINICAL TRIAL: NCT05339763
Title: Long Term Bowel Functional Outcomes Following Anal Sphincter Preserving Surgery for Rectal Cancer: A Single Center Longitudinal Study.
Brief Title: Long Term Bowel Function Following Rectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Sakr, consultant and lecturer of general surgery, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2019-1098
Record Dates: First submitted 2022-03-31; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Bowel; Functional Syndrome; Rectal Cancer
Keywords: Rectal cancer; Sphincter preserving surgery; Neoadjuvant therapy; ow anterior resection syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Rectal Neoplasms | interventions — Chemoradiotherapy; Neoadjuvant Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiation group (Active Comparator): Those are patient with rectal cancer who underwent preoperative neoadjuvant chemo radiotherapy before surgery.
  Interventions: Radiation: chemoradiotherapy
- non radiation group (Active Comparator): Those are patient with rectal cancer who did not receive preoperative neoadjuvant chemo radiotherapy before surgery.
  Interventions: Radiation: chemoradiotherapy

INTERVENTIONS:
Radiation: chemoradiotherapy — exposure of patients with rectal cancer to radiotherapy and assessment of their bowel function after surgery
  Other Names: neoadjuvant chemoradiotherapy

SUMMARY:
* In this longitudinal study, 171 patients were evaluated and compared based on the radiation therapy they received.
* Bowel function was assessed longitudinally with Memorial Sloan Kettering Cancer Center and Wexner scores every 6 months after restoration of bowel continuity. Patients with at least two follow-up visits were included.

DETAILED DESCRIPTION:
Background Despite advances in the neoadjuvant chemoradiation therapy and anal sphincter-preserving surgeries for rectal cancer, bowel dysfunction is still unavoidable which negatively affect the patients' quality of life. In this longitudinal study, The aim of this study was to investigate the changes in bowel function with follow up time and the effect of the neoadjuvant chemo radiotherapy on bowel function following low anterior resection for rectal cancer.

Materials and methods In this study, 171 patients with rectal cancer who underwent low anterior resection between 2012 and 2018 were included. Bowel function was assessed longitudinally with Memorial Sloan Kettering Cancer Center and Wexner scores every 6 months after restoration of bowel continuity. Patients with at least two follow-up visits were included.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes,
* Aged between 18 and 75 years,
* Patients with mid and upper rectal cancer (6-15) cm from the anal verge(AV) with or without preoperative chemo radiotherapy.
* Patients who underwent low anterior resection(LAR).
* Patients who were followed up with at least two outpatient visits for bowel function assessment.

Exclusion Criteria:

* Patients with recurrent rectal tumors,
* Surgically unfit patients,
* Patients with tumors infiltrating the puborectalis muscle or external sphincter.
* Patients with preoperative fecal incontinence.
* Patients who were followed up only once in the outpatient clinic.
* Patients with lower rectal cancer less than 6cm from AV,
* Patients who underwent abdominoperineal resection(APR) or intersphincteric resection(ISR).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
bowel function | 6 months-24 months
  During follow-up of the patients in the outpatient clinic, a designated nurse interviewed the patients using bowel function assessment questionnaires at different time intervals between November 2015-when bowel function assessment was started using MSKCC score-and July 2019. Each patient was interviewed at least twice.
  The Memorial Sloan Kettering Cancer Center (MSKCC) questionnaire was used. The MSKCC score questionnaire contains 18 questions divided into three subscales: the frequency subscale with six items, dietary subscale with four items, and urgency/soilage subscale with four items, with four additional single items. Each subscale is scored by adding the scores of each item, and the global score is the sum of all subscale scores. Finally, the total score is calculated by summing the global score and the scores for the four single items with the maximum score of 90. The higher the score the better the function.

SECONDARY OUTCOMES:
fecal incontinence | 6 months-24 months
  During follow-up of the patients in the outpatient clinic, a designated nurse interviewed the patients using fecal incontinence assessment questionnaire at different time intervals between November 2015-when fecal incontinence assessment was started using Wexner score-and July 2019. Each patient was interviewed at least twice.
  The Wexner questionnaire was used. Wexner score questionnaire comprises five questions regarding solid, liquid, and gas incontinence; the use of a pad; and lifestyle alterations on a scale of 0-20 (0: no incontinence; 20: complete incontinence). The lower the score, the better the continence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided